CLINICAL TRIAL: NCT00245895
Title: Phase II Study of Aranesp (Darbepoetin Alfa) to Treat Anemia in Prostate Cancer Patients.
Brief Title: Study of Aranesp to Treat Anemia in Prostate Cancer Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Amgen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 03-6503-A
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Prostate Cancer; Anemia
Keywords: Anemia,; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Aranesp
  Interventions: Drug: Aranesp

INTERVENTIONS:
Drug: Aranesp — Aranesp
  Other Names: darbepoetin

SUMMARY:
The purpose of this study is to see if darbepoetin alfa is an effective treatment for anemia in prostate cancer patients and, if so, what dose is most effective. Sometimes prostate cancer patients have low red blood cell counts (low hemoglobin) from various treatments they are receiving, such as chemotherapy. The red blood cells deliver oxygen to the tissue. This then helps give the patient more energy.

DETAILED DESCRIPTION:
This study is to evaluate the effectiveness of Darbepoetin alfa, (also referred to as Aranesp or NESP), to assess what dose of NESP is required to treat anemia in prostate cancer patients, what the side effects of NESP are, and whether NESP will affect the patients' quality of life. NESP is approved by the FDA for the treatment of anemia in patients with chronic kidney failure and for the treatment of anemia in cancer patients who are receiving chemotherapy. It is considered experimental for the treatment of anemia in prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have either histologically confirmed adenocarcinoma of the prostate or clinical evidence including a PSA greater than 50, with evidence of bone metastases, currently receiving either androgen suppression or chemotherapy.
* Patients on concurrent androgen deprivation treatment that consists of either orchiectomy or a GnRH agonist (Zoladex or Lupron) with or without and androgen receptor antagonist (Casodex, Nilandron, or Eulexin) therapy, as long as therapy was initiated within the last 3 months. Finasteride treatment must be discontinued. Secondary hormonal therapy with DES or ketoconazole is permitted.
* Patients may have a history of radiation therapy, providing that at least 6 weeks have elapsed from the last treatment date to study day 1.
* Patients must have a life expectancy of at least 12 months and a zubrod performance status of 0-2.
* Patients must not have evidence of hemolysis, and no overt gastrointestinal bleeding or bleeding due to recent surgery.
* Patients must have serum creatinine level of less than or equal to 2 mg/dL.
* Patients must have adequate liver function, as evidenced by aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2 x ULN within the 3 months prior to screening.
* Before any study-specific procedure, the patients must give written informed consent to participate in the study.

Exclusion Criteria:

* Patients presenting an active primary or metastatic malignancy involving the CNS. Patients with a previous history of primary or metastatic malignancy involving the CNS will be eligible for the study, if they have had no clinical signs or symptoms of, not treatment for CNS disease, and no history of seizures within the previous 2 years.
* Patients receiving rHuEPO therapy within 4 weeks prior to first dose of the study drug.
* Active bleeding or RBC transfusion within 4 weeks prior to fist dose of study drug.
* Patients with an active seizure disorder. Patients with a previous history of seizure disorder will be eligible for the study, if they have had no evidence of seizure activity, and they have been free of anti-convulsant medication for the previous 5 years.
* Patients with uncontrolled angina, congestive heart failure or uncontrolled cardiac arrhythmia.
* Patients with uncontrolled hypertension
* Patients with a history of hyperviscosity syndrome
* Patients with evidence of clinically significant systemic active infection or inflammatory disease
* Patients with known positive test for human immunodeficiency virus (HIV) infection
* Patients with inadequate iron stores (Fe/TIBC less than 15% and ferritin less than 10.0 mg/L)
* Patients with a history or any primary hematologic disorder that could cause anemia
* Patients currently receiving, or not yet 30 days past receiving (prior to the first dose of study drug), other investigational agents or devices not approved in any indication by the governing regulatory authority. Note: an exception will be made for patients receiving DN-101, a new formulation of calcitriol, on an investigational study.
* Patients who have previously received Aranesp (darbepoetin alfa) within 4 weeks prior to fist dose of study drug.
* Patients with a known hypersensitivity to the active substance or any of the excipients.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-04; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Hemoglobin greater than or equal to 12.5 | Feb 2005

SECONDARY OUTCOMES:
The median time to achieving the primary endpoint. | Feb 2005
The dose required to achieve the primary endpoint of more than 50% of patients. | Feb 2005
A description of the qualitative and quantitative toxicities of the administration of Aranesp (darbepoetin alfa) in this patient population. | Feb 2005
Changes in QOL from baseline compared to 3 and 6 month time point using the anemia subscale of FACT-P. | Feb 2005

CONTACTS AND LOCATIONS:
Overall Officials: Celestia S Higano, MD, Principal Investigator — University of Washington; Tomasz M Beer, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health and Sciences University, Portland, Oregon
  - Seattle Cancer Care Alliance, Seattle, Washington